CLINICAL TRIAL: NCT02352948
Title: A Phase III, Open Label, Randomised, Multi-centre, International Study of MEDI4736, Given as Monotherapy or in Combination With Tremelimumab Determined by PD-L1 Expression Versus Standard of Care in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Stage IIIB-IV) Who Have Received at Least Two Prior Systemic Treatment Regimens Including One Platinum Based Chemotherapy Regimen and Do Not Have Known EGFR TK Activating Mutations or ALK Rearrangements (ARCTIC).
Brief Title: A Global Study to Assess the Effects of MEDI4736 (Durvalumab), Given as Monotherapy or in Combination With Tremelimumab Determined by PD-L1 Expression Versus Standard of Care in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer
Acronym: ARCTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00004; 2014-000338-46 (EudraCT Number)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Non - Small Cell Lung Cancer NSCLC
MeSH Terms: interventions — durvalumab; Vinorelbine; Gemcitabine; Erlotinib Hydrochloride; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MEDI4736 (durvalumab) monotherapy in Sub-study A (Experimental): MEDI4736 (durvalumab) by intravenous infusion. Sub-study A for patients with PD-L1 positive tumors.
  Interventions: Drug: MEDI4736 (durvalumab)
- Standard of Care in Sub-study A (Active Comparator): Investigator choice from Vinorelbine, Gemcitabine and Erlotinib. Sub-study A for patients with PD-L1 positive tumors.
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine; Drug: Erlotinib
- MEDI4736 (durvalumab) + tremelimumab in Sub-study B (Experimental): MEDI4736 (durvalumab) by intravenous infusion and tremelimumab by intravenous infusion. Sub-study B for patients with PD-L1 negative tumors.
  Interventions: Drug: MEDI4736 (durvalumab) in combination with tremelimumab (anti-CTLA4)
- Standard of Care in Sub-study B (Active Comparator): Investigator choice from Vinorelbine, Gemcitabine and Erlotinib. Sub-study B for patients with PD-L1 negative tumors.
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine; Drug: Erlotinib
- MEDI4736 (durvalumab) monotherapy in Sub-study B (Experimental): MEDI4736 (durvalumab) by intravenous infusion. Sub-study B for patients with PD-L1 negative tumors.
  Interventions: Drug: MEDI4736 (durvalumab)
- tremelimumab in Sub-study B (Experimental): tremelimumab by intravenous infusion. Sub-study B for patients with PD-L1 negative tumors.
  Interventions: Drug: tremelimumab (anti-CTLA4)

INTERVENTIONS:
Drug: MEDI4736 (durvalumab) — MEDI4736 (durvalumab) treatment by intravenous infusion
  Arms: MEDI4736 (durvalumab) monotherapy in Sub-study A; MEDI4736 (durvalumab) monotherapy in Sub-study B
Drug: Vinorelbine — Vinorelbine by intravenous infusion. Administered at a dose of 30 mg/m2 iv on Days 1, 8, 15 and 22 of a 28-day cycle.
  Arms: Standard of Care in Sub-study A; Standard of Care in Sub-study B
Drug: Gemcitabine — Gemcitabine by intravenous infusion. Administered at a dose of 1000 mg/m2 iv over 30 minutes on Days 1, 8, and 15 of a 28-day cycle.
  Arms: Standard of Care in Sub-study A; Standard of Care in Sub-study B
Drug: Erlotinib — Erlotinib administered at a dose of 150 mg once daily as a tablet for oral administration
  Arms: Standard of Care in Sub-study A; Standard of Care in Sub-study B
Drug: MEDI4736 (durvalumab) in combination with tremelimumab (anti-CTLA4) — MEDI4736 (durvalumab) in combination with tremelimumab (anti-CTLA4) treatment by intravenous infusion
  Arms: MEDI4736 (durvalumab) + tremelimumab in Sub-study B
Drug: tremelimumab (anti-CTLA4) — tremelimumab (anti-CTLA4) treatment by intravenous infusion
  Arms: tremelimumab in Sub-study B

SUMMARY:
This study is a Phase III, randomised, open label, multi-centre study assessing the efficacy and safety of MEDI4736 (durvalumab) versus Standard of Care in NSCLC patients with PD-L1 positive tumours and the combination of MEDI4736 (durvalumab) plus tremelimumab (MEDI4736+treme) versus Standard of Care in NSCLC patients with PD-L1-negative tumours in the treatment of male and female patients with locally advanced or metastatic NSCLC (Stage IIIB-IV), who have received at least 2 prior systemic treatment regimens including 1 platinum-based chemotherapy regimen for NSCLC. Patients with known EGFR (Epidermal growth factor receptor) tyrosine kinase (TK) activating mutations and anaplastic lymphoma kinase (ALK) rearrangements are not eligible for the study (prospective testing is not planned within this study). The Standard of Care options are: an EGFR tyrosine kinase inhibitor (erlotinib [TARCEVA®]), gemcitabine or vinorelbine (NAVELBINE®)

DETAILED DESCRIPTION:
The study has an umbrella design with 2 sub-studies: sub-study A (randomizing patients with PD-L1 positive tumours 1:1 into MEDI4736 (durvalumab) vs. Standard of Care) and sub-study B (randomizing patients with PD-L1 negative tumours 2:3:1:2 into MEDI4736 (durvalumab) vs. MEDI4736 (durvalumab) plus tremelimumab vs. tremelimumab vs. Standard of Care. The two substudies may have different durations of recruitment periods due to differences in patient population (PD-L1 expression). They may not run concurrently with start and completion of recruitment potentially occurring at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* Documented evidence of NSCLC (Stage IIIB/ IV disease)
* Disease progression or recurrence after both a platinum-based chemotherapy regimen and at least 1 additional regimen for treatment of NSCLC
* World Health Organization (WHO) Performance Status of 0 or 1
* Estimated life expectancy more than 12 weeks

Exclusion Criteria:

* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody or anti-CTLA4
* Brain metastases or spinal cord compression unless asymptomatic, treated and stable (not requiring steroids)
* Active or prior documented autoimmune disease within the past 2 years
* Evidence of severe or uncontrolled systemic disease, including active bleeding diatheses or active infections including hepatitis B, C and HIV
* Any unresolved toxicity CTCAE (Common Terminology Criteria of Adverse Events) >Grade 2 from previous anti-cancer therapy
* Known EGFR TK activating mutations or ALK rearrangements
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, MBChB, PhD, Study Director — AstraZeneca
Locations (165):
- United States (32):
  - Research Site, Chandler, Arizona
  - Research Site, Anaheim, California
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, San Diego, California
  - Research Site, Aurora, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Waterloo, Iowa
  - Research Site, Ashland, Kentucky
  - Research Site, Rockville, Maryland
  - Research Site, Battle Creek, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, West Chester, Ohio
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Spokane, Washington
- Australia (2):
  - Research Site, Murdoch
  - Research Site, Port Macquarie
- Belgium (6):
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Libramont-Chevigny
  - Research Site, Mons
  - Research Site, Roeselare
  - Research Site, Yvoir
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Sofia
  - Research Site, Varna
- Canada (2):
  - Research Site, Moncton, New Brunswick
  - Research Site, Saint John, New Brunswick
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- Czechia (2):
  - Research Site, Nová Ves pod Pleší
  - Research Site, Prague
- France (12):
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Le Mans
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Pau
  - Research Site, Saint-Herblain
  - Research Site, Toulon
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Gauting
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Homburg
  - Research Site, Löwenstein
  - Research Site, Regensburg
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Villingen-Schwenningen
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Hungary (3):
  - Research Site, Miskolc
  - Research Site, Törökbálint
  - Research Site, Zalaegerszeg
- Research Site, Tel Litwinsky, Israel
- Italy (14):
  - Research Site, Aviano
  - Research Site, Candiolo
  - Research Site, Catania
  - Research Site, Cremona
  - Research Site, Genova
  - Research Site, Lucca
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Rimini
  - Research Site, Terni
- Japan (23):
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kobe
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Research Site, Amsterdam, Netherlands
- Poland (3):
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
- Romania (6):
  - Research Site, Alba Iulia
  - Research Site, Baia Mare
  - Research Site, Cluj-Napoca
  - Research Site, Onești
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (3):
  - Research Site, Arkhangelsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Gornji Matejevac
  - Research Site, Kamenitz
  - Research Site, Kragujevac
- Research Site, Singapore, Singapore
- South Korea (6):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Jeonnam
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (10):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Girona
  - Research Site, Jaén
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Muang
  - Research Site, Phitsanulok
  - Research Site, Songkhla
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Southampton
  - Research Site, Stevenage
  - Research Site, Truro
  - Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Martin ML, Correll J, Walding A, Ryden A. How patients being treated for non-small cell lung cancer value treatment benefit despite side effects. Qual Life Res. 2022 Jan;31(1):135-146. doi: 10.1007/s11136-021-02882-6. Epub 2021 May 31. PMID 34056687
- [Derived] Planchard D, Reinmuth N, Orlov S, Fischer JR, Sugawara S, Mandziuk S, Marquez-Medina D, Novello S, Takeda Y, Soo R, Park K, McCleod M, Geater SL, Powell M, May R, Scheuring U, Stockman P, Kowalski D. ARCTIC: durvalumab with or without tremelimumab as third-line or later treatment of metastatic non-small-cell lung cancer. Ann Oncol. 2020 May;31(5):609-618. doi: 10.1016/j.annonc.2020.02.006. Epub 2020 Feb 20. PMID 32201234
- See also: AstraZeneca Cancer Study Locator Service astrazeneca@emergingmed.com Phone number: 1-877-400-465 — http://www.emergingmed.com/networks/AstraZeneca
- See also: Redacted SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2584&filename=D4191C00004-sap-arctic-ed-3_Redacted.pdf
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2584&filename=D4191C00004-revised-csp-7_Redacted.pdf
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191C00004&attachmentIdentifier=6739cb21-2029-418c-8f56-df0682607b8b&fileName=d4191c00004-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was divided into 2 parts, sub-study A (82 centers across Europe, Asia, and North America) and sub-study B (149 centers across Europe, Asia, North America, and South America) conducted between 13 January 2015 and 09 February 2018 (data cut-off date).
Pre-assignment Details: The study had a pre-screening period to determine the programmed cell death ligand 1 (PD-L1) status, followed by a screening period and 12 month treatment period. A total of 595 participants were randomized to either sub-study A [PD-L1 high (>=25% of tumor cell (TC) expressing PD-L1)] or sub-study B [PD-L1 low/neg (<25% of TC expressing PD-L1)].
Groups:
- Sub-study A: Durvalumab: Participants received durvalumab (MEDI4736) 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks (Q2W) for 12 months (up to 26 doses).
- Sub-study A: Standard of Care (SoC): Participants received either erlotinib 150 mg tablet orally once daily; gemcitabine 1000 mg/meter square (m^2) IV infusion on Days 1, 8, and 15 of a 28-day cycle; or vinorelbine 30 mg/m^2 IV infusion on Days 1, 8, 15, and 22 of a 28-day cycle until progression of disease (PD), initiation of alternative anti-cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment criterion occurred.
- Sub-study B: Durvalumab+Tremelimumab: Participants received durvalumab 20 mg/kg plus tremelimumab 1 mg/kg IV infusion every 4 weeks (Q4W) for 12 weeks (4 doses) followed by durvalumab alone 10 mg/kg IV infusion Q2W for 34 weeks starting at Week 16 (up to 18 additional doses).
- Sub-study B: SoC: Participants received either erlotinib 150 mg tablet orally once daily; gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of a 28-day cycle; or vinorelbine 30 mg/m^2 IV infusion on Days 1, 8, 15, and 22 of a 28-day cycle until PD, initiation of alternative anti-cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment criterion occurred.
- Sub-study B: Durvalumab: Participants received durvalumab 10 mg/kg IV infusion Q2W for 12 months (up to 26 doses).
- Sub-study B: Tremelimumab: Participants received tremelimumab 10 mg/kg IV infusion Q4W for 24 weeks followed by every 12 weeks (Q12W) for 24 weeks (up to 9 doses).
Period: Overall Study
Arm/Group | Sub-study A: Durvalumab | Sub-study A: Standard of Care (SoC) | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Started | 62 | 64 | 174 | 118 | 117 | 60
Received Treatment | 62 | 63 | 173 | 110 | 117 | 60
Completed Study Treatment | 15 | 0 | 36 | 0 | 23 | 4
Completed (Completed the Study) | 13 | 5 | 45 | 19 | 29 | 11
Not Completed | 49 | 59 | 129 | 99 | 88 | 49
Not completed — Death | 47 | 48 | 114 | 74 | 77 | 44
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 10 | 11 | 23 | 9 | 4
Not completed — Eligibility criteria not fulfilled | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sub-study A and B: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Groups:
- Sub-study A: Durvalumab; Sub-study B: Durvalumab: Participants received durvalumab 10 mg/kg IV infusion Q2W for 12 months (up to 26 doses).
- Sub-study A: SoC; Sub-study B: SoC: Participants received either erlotinib 150 mg tablet orally once daily; gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of a 28-day cycle; or vinorelbine 30 mg/m^2 IV infusion on Days 1, 8, 15, and 22 of a 28-day cycle until PD, initiation of alternative anti-cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment criterion occurred.
- Sub-study B: Durvalumab+Tremelimumab: Participants received durvalumab 20 mg/kg plus tremelimumab 1 mg/kg IV infusion Q4W for 12 weeks (4 doses) followed by durvalumab alone 10 mg/kg IV infusion Q2W for 34 weeks starting at Week 16 (up to 18 additional doses).
- Sub-study B: Tremelimumab: Participants received tremelimumab 10 mg/kg IV infusion Q4W for 24 weeks followed by Q12W for 24 weeks (up to 9 doses).
- Total: Total of all reporting groups
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab | Total
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60 | 595
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 3 | 11 | 16 | 8 | 13 | 4 | 55
  >=50 to <65 years | 31 | 25 | 79 | 49 | 52 | 27 | 263
  >=65 to <75 years | 24 | 21 | 64 | 50 | 39 | 24 | 222
  >=75 years | 4 | 7 | 15 | 11 | 13 | 5 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 59 | 37 | 44 | 21 | 197
  Male | 42 | 48 | 115 | 81 | 73 | 39 | 398
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 22 | 23 | 41 | 41 | 34 | 16 | 177
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 2 | 2 | 1 | 9
  White | 40 | 40 | 129 | 74 | 79 | 43 | 405
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From randomization (Day 1) until death due to any cause, approximately 36 months
Population: Sub-study A and B: FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC
Number analyzed (Participants) | 62 | 64 | 174 | 118
months | 11.7 [8.2 to 17.4] | 6.8 [4.9 to 10.2] | 11.5 [8.7 to 14.1] | 8.7 [6.5 to 11.7]
Statistical Analysis 1: Comparison: Sub-study A: Durvalumab vs Sub-study A: SoC; For sub-study A: durvalumab monotherapy treatment arm was compared with SoC; Test type: Other — Sub-study A was not powered and thus no formal statistical comparisons were performed; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.42 to 0.93] — Hazard ratio and CI are estimated from a stratified Cox proportional hazards model with Breslow method to control for ties, stratification factors SoC therapy, and histology in strata statement, and CI is calculated using profile likelihood approach
Statistical Analysis 2: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: SoC; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with SoC; Test type: Superiority; p = 0.109, Log Rank; The P-value arises from a stratified log-rank test adjusting for SoC therapy and histology, with ties handled by the Breslow approach; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.61 to 1.05] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression. The PFS was determined by Investigator assessments according to response evaluation criteria in solid tumours (RECIST) version 1.1. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 millimeter (mm) or progression of non-target lesions or the appearance of a new lesion
Time Frame: Tumour scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed up to a maximum of approximately 3 years.
Population: Sub-study A and B: FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC
Number analyzed (Participants) | 62 | 64 | 174 | 118
months | 3.8 [1.9 to 5.6] | 2.2 [1.9 to 3.7] | 3.5 [2.3 to 4.6] | 3.5 [1.9 to 3.9]
Statistical Analysis 1: Comparison: Sub-study A: Durvalumab vs Sub-study A: SoC; For sub-study A: durvalumab monotherapy treatment arm was compared with SoC; Test type: Other — Sub-study A was not powered and thus no formal statistical comparisons were performed; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.49 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: SoC; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with SoC; Test type: Superiority; p = 0.056, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.59 to 1.01] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: OS, Contribution of the Components Analysis of Sub-study B
Description: The OS was defined as the time from the date of randomization until death due to any cause.
Time Frame: From randomization (Day 1) until death due to any cause, approximately 36 months
Population: FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 174 | 117 | 60
months | 11.5 [8.7 to 14.1] | 10.0 [7.1 to 13.2] | 6.9 [3.9 to 13.2]
Statistical Analysis 1: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Durvalumab; As part of the contribution of components analysis for sub-study B, durvalumab plus tremelimumab treatment arm was compared with durvalumab monotherapy; Test type: Superiority; p = 0.885, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.74 to 1.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Tremelimumab; As part of the contribution of components analysis for sub-study B, durvalumab plus tremelimumab treatment arm was compared with tremelimumab monotherapy; Test type: Superiority; p = 0.153, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.56 to 1.11] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Alive at 12 Months (OS12)
Description: The OS12 was defined as the percentage of participants who were alive at 12 months after randomisation per Kaplan-Meier estimate of OS at 12 months.
Time Frame: From randomization (Day 1) up to 12 months
Population: Sub-study A and B: FAS included all randomized participants analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60
percentage of participants | 49.3 [36.3 to 61.0] | 31.3 [20.2 to 43.0] | 49.5 [41.7 to 56.7] | 38.8 [29.9 to 47.7] | 43.6 [34.4 to 52.4] | 41.2 [28.7 to 53.3]
Statistical Analysis 1: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: SoC; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with SoC; Test type: Superiority; p = 0.063, z-test — The z-test statistic is the ratio of log-transformed ratio of the cumulative hazards in the 2 treatment arms divided by square root of the variance; The variance is estimated using the delta method and Greenwood's formula

5. Secondary Outcome: PFS, Contribution of the Components Analysis of Sub-study B
Description: The PFS was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression. The PFS was determined by Investigator assessments according to RECIST v1.1. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 millimeter (mm) or progression of non-target lesions or the appearance of a new lesion
Time Frame: as for outcome 2
Population: FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 174 | 117 | 60
months | 3.5 [2.3 to 4.6] | 3.1 [1.9 to 3.7] | 2.1 [1.8 to 3.2]
Statistical Analysis 1: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Durvalumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.282, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.68 to 1.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Tremelimumab; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.011, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.92] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with at least 1 visit response of complete response (CR) or partial response (PR) among ITT participants who had measurable disease at baseline. CR was defined as disappearance of all target lesions (any pathological lymph nodes selected as target lesions must have a reduction in short axis to <10 mm) and PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum of diameters as long as criteria for PD are not met). The ORR was measured using Investigator assessments according to RECIST v1.1.
Time Frame: as for outcome 2
Population: Sub-study A and B: FAS included all randomized participants with measureable disease at baseline analyzed on an ITT basis.
Measure: Number; unit: percentage of participants
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60
percentage of participants | 35.5 | 12.5 | 14.9 | 6.8 | 15.4 | 6.7
Statistical Analysis 1: Comparison: Sub-study A: Durvalumab vs Sub-study A: SoC; For sub-study A: durvalumab monotherapy treatment arm was compared with SoC; Test type: Other — Sub-study A was not powered and thus no formal statistical comparisons were performed; Odds Ratio (OR) = 3.87, 95% CI 2-sided [1.61 to 10.10] — The analysis was performed using logistic regression adjusting for SoC therapy (gemcitabine/vinorelbine versus erlotinib) and histology (squamous versus all other histology types), with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: SoC; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with SoC; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.10 to 5.94] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Durvalumab; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with durvalumab monotherapy; Test type: Superiority; p = 0.923, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.51 to 1.89] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: Tremelimumab; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with tremelimumab monotherapy; Test type: Superiority; p = 0.109, Regression, Logistic; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.91 to 8.61] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Duration of Response (DoR)
Description: The DoR was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The DoR was determined by Investigator assessments according to RECIST v1.1. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 millimeter (mm) or progression of non-target lesions or the appearance of a new lesion
Time Frame: as for outcome 2
Population: Sub-study A and B: FAS included all randomized participants with measureable disease at baseline analyzed on an ITT basis. Only participants with objective response were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60
months | 9.5 [3.0 to 17.8] | 4.8 [1.9 to 7.6] | 12.2 [6.5 to NA] — The upper limit of the 75th percentile was not calculated as it was not reached. | 10.8 [5.6 to 12.2] | 10.0 [4.0 to NA] — The upper limit of the 75th percentile was not calculated as it was not reached. | 4.7 [2.9 to NA] — The upper limit of the 75th percentile was not calculated as it was not reached.

8. Secondary Outcome: Percentage of Participants Alive and Progression Free at 6 Months (APF6)
Description: The APF6 was defined as the percentage of participants who were alive and progression free per RECIST v1.1 at 6 months after randomization per Kaplan-Meier estimate of PFS at 6 months. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 millimeter (mm) or progression of non-target lesions or the appearance of a new lesion
Time Frame: Tumour scans performed at baseline then every ~8 weeks up to 6 months
Population: Sub-study A and B: FAS included all randomized participants analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60
percentage of participants | 35.5 [23.9 to 47.3] | 24.1 [14.1 to 35.6] | 31.5 [24.6 to 38.7] | 27.6 [19.0 to 36.7] | 27.2 [19.4 to 35.6] | 14.5 [6.9 to 24.9]

9. Secondary Outcome: Percentage of Participants Alive and Progression Free at 12 Months (APF12)
Description: The APF12 was defined as the percentage of participants who were alive and progression free per RECIST v1.1 at 12 months after randomization per Kaplan-Meier estimate of PFS at 12 months. PD was defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 millimeter (mm) or progression of non-target lesions or the appearance of a new lesion
Time Frame: Tumour scans performed at baseline then every ~8 weeks up to 12 months.
Population: Sub-study A and B: FAS included all randomized participants analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 62 | 64 | 174 | 118 | 117 | 60
percentage of participants | 19.4 [10.7 to 30.0] | 9.9 [3.8 to 19.3] | 20.6 [14.7 to 27.1] | 8.0 [3.4 to 15.2] | 15.0 [9.1 to 22.3] | 7.3 [2.4 to 16.0]

10. Secondary Outcome: Time From Randomisation to Second Progression (PFS2) of Sub-study B
Description: The PFS2 was defined as the time from the date of randomization to the earliest of the progression event subsequent to that used for the PFS endpoint or death and determined by local standard clinical practice and have included any of the following: objective radiological, symptomatic progression, or death. PFS2 was reported for sub-study B only.
Time Frame: Tumour scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~12 weeks thereafter until first progression. Disease then assessed per local practice until 2nd progression. Assessed up to a maximum of approximately 3 years.
Population: FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
Number analyzed (Participants) | 174 | 118 | 117 | 60
months | 9.1 [6.6 to 12.3] | 6.7 [4.7 to 8.9] | 8.0 [6.3 to 10.0] | 5.7 [3.2 to 10.0]
Statistical Analysis 1: Comparison: Sub-study B: Durvalumab+Tremelimumab vs Sub-study B: SoC; For sub-study B: durvalumab plus tremelimumab treatment arm was compared with SoC; Test type: Superiority; p = 0.002, Log Rank; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.85] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From signature of informed consent up to 90 days after the last dose of durvalumab and/or tremelimumab and 30 days after the last dose of SoC, approximately 15 months.
Description: Sub-study A and B: Safety analysis set included all participants who received at least 1 dose of randomized treatment. All-cause mortality is defined as death due to any cause (including disease progression) for the entire duration of the study.
Groups:
- Sub-study A: SoC; Sub-study B: SoC: Participants received either erlotinib 150 mg tablet orally once daily; gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of a 28-day cycle; or vinorelbine 30 mg/m^2 IV infusion on Days 1, 8, 15, and 22 of a 28-day cycle until PD, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment criterion occurred.
Arm/Group | Sub-study A: Durvalumab | Sub-study A: SoC | Sub-study B: Durvalumab+Tremelimumab | Sub-study B: SoC | Sub-study B: Durvalumab | Sub-study B: Tremelimumab
All-Cause Mortality (participants affected / at risk) | 48/62 | 55/64 | 118/174 | 90/118 | 83/117 | 46/60
Serious Adverse Events (participants affected / at risk) | 23/62 | 16/63 | 65/173 | 28/110 | 36/117 | 23/60
Other Adverse Events (participants affected / at risk) | 52/62 | 59/63 | 139/173 | 100/110 | 99/117 | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-study A: Durvalumab (N=62) | Sub-study A: SoC (N=63) | Sub-study B: Durvalumab+Tremelimumab (N=173) | Sub-study B: SoC (N=110) | Sub-study B: Durvalumab (N=117) | Sub-study B: Tremelimumab (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perforation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 3 (3) | 7 (7) | 2 (2) | 2 (2) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (7) | 2 (2) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-study A: Durvalumab (N=62) | Sub-study A: SoC (N=63) | Sub-study B: Durvalumab+Tremelimumab (N=173) | Sub-study B: SoC (N=110) | Sub-study B: Durvalumab (N=117) | Sub-study B: Tremelimumab (N=60)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 17 (22) | 17 (18) | 27 (49) | 11 (13) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (8) | 2 (3) | 7 (15) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (40) | 3 (7) | 18 (48) | 0 (0) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 5 (10) | 3 (6) | 11 (15) | 4 (4) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 17 (17) | 0 (0) | 6 (7) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (6) | 0 (0) | 14 (15) | 1 (1) | 10 (11) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4) | 5 (5) | 2 (5) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (6) | 7 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (15) | 15 (16) | 14 (15) | 11 (12) | 15 (16) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 8 (8) | 36 (45) | 18 (26) | 25 (33) | 16 (20)
Nausea (Gastrointestinal disorders) | 11 (12) | 15 (20) | 28 (33) | 22 (32) | 20 (25) | 11 (16)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 5 (5) | 10 (11) | 5 (6) | 3 (3) | 1 (3)
Vomiting (Gastrointestinal disorders) | 8 (8) | 4 (5) | 17 (17) | 8 (13) | 18 (22) | 7 (10)
Asthenia (General disorders) | 6 (6) | 8 (17) | 31 (39) | 17 (19) | 16 (21) | 9 (9)
Fatigue (General disorders) | 10 (10) | 10 (16) | 25 (27) | 24 (30) | 22 (24) | 4 (4)
Malaise (General disorders) | 1 (1) | 4 (8) | 3 (3) | 5 (5) | 8 (8) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 2 (3) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 6 (8) | 3 (5) | 16 (17) | 9 (10) | 8 (10) | 2 (3)
Pyrexia (General disorders) | 9 (14) | 6 (8) | 20 (27) | 23 (33) | 12 (15) | 6 (7)
Influenza (Infections and infestations) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (1) | 15 (18) | 5 (5) | 7 (8) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 3 (3) | 10 (11) | 10 (15) | 5 (9) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 11 (12) | 8 (12) | 2 (5) | 5 (6)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4) | 2 (3) | 3 (6) | 4 (5) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 4 (5) | 2 (3) | 4 (4) | 1 (1) | 1 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 9 (33) | 2 (2) | 18 (43) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 6 (8) | 1 (1) | 8 (27) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 6 (7) | 4 (4) | 14 (14) | 4 (4) | 8 (8) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 6 (21) | 2 (2) | 11 (32) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19) | 20 (24) | 34 (39) | 23 (24) | 27 (28) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3) | 3 (3) | 2 (2) | 8 (10) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3) | 16 (19) | 2 (4) | 10 (10) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (7) | 11 (13) | 4 (4) | 14 (15) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 7 (7) | 2 (2) | 7 (7) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 4 (4) | 7 (10) | 5 (5) | 12 (12) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 9 (9) | 4 (4) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 9 (11) | 5 (5) | 9 (11) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 9 (11) | 25 (26) | 15 (16) | 16 (17) | 6 (6)
Dizziness (Nervous system disorders) | 6 (6) | 5 (5) | 9 (10) | 5 (6) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 9 (11) | 7 (8) | 17 (19) | 6 (8) | 8 (8) | 5 (6)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4) | 6 (6) | 5 (5) | 7 (7) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 5 (5) | 24 (29) | 14 (15) | 15 (20) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 2 (2) | 6 (7) | 4 (4) | 7 (7) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (6) | 6 (11) | 4 (4) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 4 (4) | 5 (5) | 4 (6) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2) | 28 (36) | 5 (5) | 11 (12) | 14 (17)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 9 (9) | 14 (15) | 17 (17) | 7 (9) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT02352948/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT02352948/SAP_000.pdf